CLINICAL TRIAL: NCT03668288
Title: Tolerance and Patients' Satisfaction of Subcutaneous Infusion of Human Immunoglobulin Facilitated by Recombinant Human Hyaluronidase for Primary or Secondary Immunodeficiency
Brief Title: Tolerance and Patients' Satisfaction With IGHy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO18123
Record Dates: First submitted 2018-09-11; First posted 2018-09-12 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2018-09

CONDITIONS: Secondary or Primary Immunodeficiency
Keywords: IVIG; PID; home infusion; hyaluronidase; immunoglobulin; secondary and primary immunodeficiency disease; tolerance
MeSH Terms: conditions — Neoplasm Metastasis; Primary Immunodeficiency Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PID patients: Adults with primary or secondary immunodeficiency for whom human immunoglobulin-assisted recombinant human hyaluronidase treatment is initiated
  Interventions: Other: Data record and questionnaires passation

INTERVENTIONS:
Other: Data record and questionnaires passation — Data record and questionnaires passation (SF36)

SUMMARY:
Primary immunodeficiencies (PID) represent more than 150 diseases affecting the immune system. More than 50% of PIDs are due to a lack or an insufficiency in antibody production. Some of these immunodeficiencies as well as some secondary immune deficiency with deficient antibody production (especially in hematology and oncology) are responsible for repeated and/or severe infections, requiring long-term replacement therapy with intravenous polyclonal immunoglobulin. Intravenous replacement therapy is administered every 21 or 28 days in hospital. Subcutaneous administration (weekly or bi-weekly) can be initiated for patients who cannot tolerate intravenous infusions or who have difficult venous access. However, some patients experience a decrease in quality of life with these more frequent administration at home. A new treatment is available in France since 2017, which is a subcutaneous infusion of human immunoglobulin facilitated by recombinant human hyaluronidase (IGHy), administered every 3 to 4 weeks in a single abdominal site, at home. No direct data are available in adults to evaluate tolerance and satisfaction with this treatment, but we know it is a preferred option in children and adolescents.

DETAILED DESCRIPTION:
The objective of the study is to describe the continuation of the human immunoglobulin-assisted recombinant human hyaluronidase (IGHy) therapy at 6 months from the start of treatment.

The secondary objectives are to evaluate the quality of life of patients treated with human immunoglobulin-assisted recombinant human hyaluronidase (IGHy) therapy.

ELIGIBILITY:
Inclusion Criteria:

* major (> 18 years),
* with primary or secondary immunodeficiency,
* followed in the Department of Internal Medicine, Infectious Diseases - Clinical Immunology CHU Reims.
* Benefiting from human immunoglobulin treatment facilitated by recombinant human hyaluronidase,
* agreeing to participate in the study.

Exclusion Criteria:

* patients refusing to participate in the study
* minors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients over 18 years old
  * Patients with primary or secondary immunodeficiency
  * Patients for whom treatment with IGHy is in place.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-02-14 (Actual); Primary Completion 2020-08-14 (Estimated); Study Completion 2021-08-14 (Estimated)

PRIMARY OUTCOMES:
Continuation of the human immunoglobulin-assisted recombinant human hyaluronidase (IGHy) | Month 6
  Percentage of patients continuing IGHy treatment at 6 months

SECONDARY OUTCOMES:
quality of life assessed by the SF-36 | Month 6
  quality of life assessed by the SF-36. The Medical Outcomes Short-Form 36-Item Health Survey (SF-36v2) is a self-administered questionnaire comprising 36-items measuring eight dimensions of general HRQOL: physical functioning (10 items), role limitation due to physical health problems (4 items), bodily pain (2 items), general health perceptions (5 items), vitality (4 items), social functioning (2 items), role limitations due to emotional problems (3 items), and general mental health (5 items). In addition to scores for individual dimensions, two summary scores assessing physical and mental dimensions of health and well-being can also be calculated: Physical Component Summary (PCS) score and the Mental Component Summary (MCS) score, respectively

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France